CLINICAL TRIAL: NCT02383017
Title: Effects of Shroom Tech Sport Supplementation and Concurrent Training on Body Composition, Performance and Health in Collegiate-aged Men
Brief Title: Effects of Shroom Tech Sport Supplementation and Concurrent Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Michael J. Ormsbee, Associate Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Florida StateU
Record Dates: First submitted 2015-02-07; First posted 2015-03-09 (Estimated); Results first posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Body Composition; Performance Measures; Hormone Profiles; Blood Lipid Profiles
Keywords: Multi-ingredient performance supplement, High Intensity Interval Training, Concurrent training

STUDY DESIGN:
Intervention Model Description: A 12-week training model with testing weeks at baseline, mid point (week 7) and post-training.
Who Masked: Participant, Investigator
Masking Description: Double blind, placebo and supplement intervention
Oversight: Data Monitoring Committee: No

ARMS (2):
- Shroom Tech Sport (Experimental): Shroom Tech Sport is a multi-ingredient performance supplement taken, in pill form, prior to work outs to enhance workout performance.
  Interventions: Dietary Supplement: Shroom Tech Sport
- Placebo (Placebo Comparator): The placebo is a calorie matched sugar pill that will be taken in the same fashion as the STS pill.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Shroom Tech Sport — STS will be given every day in accordance to company guidelines for 12 weeks.
  Other Names: STS
  Arms: Shroom Tech Sport
Dietary Supplement: Placebo — Placebo will be given in the same fashion as the STS pills guidelines for 12 weeks.
  Arms: Placebo

SUMMARY:
This study will examine how the supplement Shroom Tech Sport (STS) affects body composition and different performance and health measures over the course of 12 weeks. The supplement will be combined with a concurrent training regime consisting of resistance and high intensity interval training. Subjects will be tested for percent body fat to determine body composition. Further, they will also be tested for maximal strength (squat and bench), maximal power output and fatigue, lactate threshold and maximal oxygen volume consumption (VO2max). And finally, subjects will be tested for health and hormone markers in the blood. All of these measures will be compared against a placebo group participating in the same exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

1. participate in the 3-4 week supplement wash out prior to beginning the experiment (except for basic protein supplements and multivitamins)
2. have at least 1 year of recreational exercise with a minimum of three times a week

Exclusion Criteria:

1. Prior steroid use
2. History of tumors
3. Pre-existing musculoskeletal disorders

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-07-30 (Actual); Study Completion 2016-07-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sports Science and Medicine, Florida State University, Tallahassee, Florida, United States

REFERENCES:
- [Derived] Kreipke PhD VC, Moffatt PhD RJ, Tanner Ma CJ, Ormsbee PhD MJ. Effects of Concurrent Training and a Multi-Ingredient Performance Supplement Containing Rhodiola rosea and Cordyceps sinensis on Body Composition, Performance, and Health in Active Men. J Diet Suppl. 2021;18(6):597-613. doi: 10.1080/19390211.2020.1822486. Epub 2020 Oct 20. PMID 33078636

RESULTS

PARTICIPANT FLOW:
Groups:
- Shroom Tech Sport: This group consumed Shroom Tech Sport in accordance with manufacturer's instructions (one pill per 23kg (50lbs)) 45 minutes prior to exercise and testing and with breakfast on non-training days.
- Placebo: This group consumed the placebo in accordance with the instructions provided for Shroom Tech Sport. Participants consumed one pill per 23kg (50lbs) 45 minutes before exercise and testing and with breakfast on non-training days.
Period: Overall Study
Arm/Group | Shroom Tech Sport | Placebo
Started | 15 | 13
Completed | 10 | 11
Not Completed | 5 | 2
Not completed — Injury Sustained Outside Study | 1 | 0
Not completed — Compliance | 3 | 2
Not completed — Found to be Hypogonadal | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Shroom Tech Sport | Placebo | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 21.5 (1.2) | 22.5 (2.7) | 22 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 11 | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 21
Height [Mean (Standard Deviation); unit: cm] | 176.4 (7.2) | 175.9 (3.4) | 176.2 (5.3)
Weight [Mean (Standard Deviation); unit: kg] | 75.4 (8.1) | 76 (8.8) | 75.7 (8.5)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.2 (1.8) | 24.6 (2.7) | 24.4 (2.3)
Years of Prior Training Experience [Mean (Standard Deviation); unit: years] — This is the number of years of training experience that the participants had before entering the study
  years | 6.4 (2.8) | 5.8 (2.7) | 6.1 (2.8)
Percentage of Body Fat [Mean (Standard Deviation); unit: Percent] — Percent of total weight that is body fat weight
  Percent | 15.5 (5.8) | 16.2 (6.7) | 15.9 (6.3)
Total Strength [Mean (Standard Deviation); unit: kg] — This is the sum of the two tested lifts, bench and squat
  kg | 223 (29) | 217 (40) | 220 (35)
VO2max (ml/kg/min) [Mean (Standard Deviation); unit: ml/kg/min] | 54.3 (6.7) | 54.3 (5.7) | 54.3 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Fat as Measured by Bod Pod
Description: Changes in percent body fat
Time Frame: Baseline,Week 7, Week 14
Measure: Mean (Standard Deviation); unit: Percent Body Fat
Arm/Group | Shroom Tech Sport | Placebo
Number analyzed (Participants) | 10 | 11
Percent Body Fat
  Baseline | 15.5 (5.8) | 16.2 (6.7)
  Week 7 | 14.8 (7.2) | 15.3 (6.5)
  Week 14 | 14.2 (6.6) | 14.3 (6.4)

2. Primary Outcome: Change in Strength as Measured by Bench and Squat One Repetition Maximum
Description: Changes in strength measures for both bench press and back squat
Time Frame: Baseline, Week 7, Week 14
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Shroom Tech Sport | Placebo
Number analyzed (Participants) | 10 | 11
kg
  Baseline | 223 (29) | 217 (40)
  Week 7 | 222 (29) | 222 (39)
  Week 14 | 234 (28) | 232 (49)

3. Primary Outcome: Change in Maximum Oxygen Consumption as Measured by VO2max Treadmill Protocol
Description: Changes in maximal oxygen consumption
Time Frame: Baseline,Week 7,Week 14
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Shroom Tech Sport | Placebo
Number analyzed (Participants) | 10 | 11
ml/kg/min
  Baseline | 54.3 (6.7) | 54.3 (5.7)
  Week 7 | 55.7 (6.4) | 56.0 (6.0)
  Week 14 | 56.5 (4.8) | 55.7 (5.7)

4. Primary Outcome: Change in Serum Hormone Concentrations
Description: Changes in Testosterone levels
Time Frame: Baseline,Week 7,Week 14
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Shroom Tech Sport | Placebo
Number analyzed (Participants) | 10 | 11
ng/ml
  Baseline | 5.9 (1.1) | 5.8 (1.2)
  Week 7 | 5.2 (1.1) | 5.7 (1.6)
  Week 14 | 5.0 (1.8) | 5.7 (1.4)

5. Primary Outcome: Change in Serum Hormone Concentrations
Description: Changes in Cortisol Levels
Time Frame: Baseline,Week 7,Week 14
Measure: Mean (Standard Deviation); unit: ug/dL
Arm/Group | Shroom Tech Sport | Placebo
Number analyzed (Participants) | 10 | 11
ug/dL
  Baseline | 19.7 (5.2) | 17.6 (4.6)
  Week 7 | 18.7 (4.2) | 17.9 (6.1)
  Week 14 | 16.4 (4.5) | 16.6 (4.3)

6. Primary Outcome: Change in Serum Hormone Concentrations
Description: Changes in IGF-I Levels
Time Frame: Baseline, Week 7, Week 14
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Shroom Tech Sport | Placebo
Number analyzed (Participants) | 10 | 11
ng/ml
  Baseline | 87.3 (22.8) | 83.9 (19.1)
  Week 7 | 92.4 (15.5) | 82.6 (21.4)
  Week 14 | 94.1 (27.1) | 80.3 (20.8)

7. Primary Outcome: Change in Serum Hormone Concentrations
Description: Changes in Sex Hormone Binding Globulin Levels
Time Frame: Baseline, Week 7, Week 14
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Shroom Tech Sport | Placebo
Number analyzed (Participants) | 10 | 11
nmol/L
  Baseline | 27.0 (6.7) | 29.0 (14.2)
  Week 7 | 29.0 (11.8) | 30.6 (17.3)
  Week 14 | 28.5 (7.7) | 29.2 (14.2)

8. Primary Outcome: Change in Strength as Measured by Bench One Repetition Maximum
Description: Changes in strength measures for bench press
Time Frame: Baseline, Week 7, Week 14
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Shroom Tech Sport | Placebo
Number analyzed (Participants) | 10 | 11
kg
  Baseline | 100 (14) | 100 (20)
  Week 7 | 98 (12) | 100 (19)
  Week 14 | 102 (14) | 105 (18)

9. Primary Outcome: Change in Strength as Measured by Squat One Repetition Maximum
Description: Changes in strength measures for Squat
Time Frame: Baseline, Week 7, Week 14
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Shroom Tech Sport | Placebo
Number analyzed (Participants) | 10 | 11
kg
  Baseline | 123 (16) | 118 (22)
  Week 7 | 128 (16) | 123 (22)
  Week 14 | 132 (15) | 128 (24)

ADVERSE EVENTS:
Arm/Group | Shroom Tech Sport | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 1/10 | 2/11
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Shroom Tech Sport (N=10) | Placebo (N=11)
Headache (General disorders) | 0 (0) | 1 (1)
Dry Mouth (General disorders) | 0 (0) | 1 (1)
Difficulty Sleeping (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No